CLINICAL TRIAL: NCT05215379
Title: Multicenter Prospective Randomized Clinical Trial of Neoadjuvant Chemoradiation Therapy Combined With Immunotherapy for MSS Ultra-low Rectal Cancer
Brief Title: Neoadjuvant Chemoradiation Therapy Combined With Immunotherapy for MSS Ultra-low Rectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Chief physician, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHCRS-Immunity
Record Dates: First submitted 2022-01-05; First posted 2022-01-31 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Neoadjuvant Chemoradiation Therapy; Rectal Cancer; Immunotherapy; Microsatellite Instability Low
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant chemoradiation therapy (Other): neoadjuvant chemoradiation therapy
  Interventions: Other: Control
- neoadjuvant chemoradiation therapy +immunotherapy (Experimental): neoadjuvant chemoradiation therapy +immunotherapy
  Interventions: Drug: xintilimab injection

INTERVENTIONS:
Drug: xintilimab injection — neoadjuvant chemoradiation therapy +xintilimab injection 200mg/3week 4cycle
  Arms: neoadjuvant chemoradiation therapy +immunotherapy
Other: Control — neoadjuvant chemoradiation therapy
  Arms: neoadjuvant chemoradiation therapy

SUMMARY:
At present, there are no relevant studies or reports on the effect of neoadjuvant chemoradiation therapy combined with immunotherapy for MSS ultra-low rectal cancer. Studied in this paper combin neoadjuvant chemoradiation with immune therapy, carry out "Multicenter prospective randomized clinical trial of neoadjuvant chemoradiation therapy combined with immunotherapy for MSS ultra-low rectal cancer" in order to provide a high-level evidence-based medical evidence for ultra-low rectal cancer treatment and improve ultra-low rectal cancer diagnosis and treatment effect.

ELIGIBILITY:
Inclusion Criteria:

Ultra low rectal cancer patients evaluated by multidisciplinary team to perform APR

* Patients who have a strong desire to preserve the anus and are willing to accept neoadjuvant treatment
* 18 years old ≤ age ≤ 75 years old, no gender limit;
* Colonoscopy, intracavitary ultrasound and pelvic high-resolution MRI (or enhanced CT) were diagnosed as extremely low rectal cancer within 5 cm from the lower edge of the tumor to the anal edge. The baseline clinical stage is T1-3aN0-1M0, and the size of the tumor <1/2 circle;
* Histopathological diagnosis of rectal adenocarcinoma; tumor biopsy immunohistochemistry showed pMMR, that is, MSH1, MSH2, MSH6 and PMS2 four proteins are positive, or genetic testing suggests MSI-L or MSS.
* The patient has good compliance and can come to the hospital for reexamination as required;
* ECOG physical status score 0-1 points;
* Have not received anti-tumor and immunotherapy before being selected;
* 8. Laboratory inspections must meet the following standards: i. White blood cell count ≥3.5×109/L, absolute neutrophil count ≥1.8×109/L, platelet count ≥100×10^9/L, hemoglobin ≥100g/L; ii. INR≤1.5, and APTT≤1.5 times the upper limit of normal value or partial prothrombin time (PTT)≤1.5 times the upper limit of normal value; iii. Total bilirubin≤1.25 times the upper limit of normal; ALT and AST≤5 times the upper limit of normal; iv. 24h creatinine clearance rate ≥50mL/min or blood creatinine ≤1.5 times the upper limit of normal.
* Voluntarily sign the informed consent form;

Exclusion Criteria:

* History of other malignant diseases in the past 5 years;
* Patients with metastases ;
* Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. who need emergency surgery;
* Those who are known to be allergic to capecitabine, oxaliplatin, PD-1 monoclonal antibody and other drugs;
* Patients with poorly differentiated adenocarcinoma, signet ring cell carcinoma, and mucinous adenocarcinoma;
* The patient is accompanied by any unstable systemic diseases, including but not limited to: severe infection, uncontrolled diabetes, hypertension that cannot be controlled by drugs, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardium Infarction, congestive heart failure, severe arrhythmia requiring medication, liver, kidney or metabolic diseases; diseases that affect the life of the patient.
* The patient's accompanying diseases (such as mental illness, etc.) or conditions (such as alcohol or drug abuse, etc.) will increase the patient's risk of receiving experimental drug treatment or affect the patient's compliance with the trial requirements, or may confuse the research results;
* Within 30 days before screening, the patient has received any other experimental drug treatment or participated in another interventional clinical trial;
* Women who are pregnant or breastfeeding or who intend to become pregnant or breastfeeding during the study period; men or women who are unwilling to take effective contraceptive measures;
* The investigator judges that the patient is not suitable to participate in other situations such as the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
The rate of cCR | 2 years
  Rate of patients who achieve clinical complete response

SECONDARY OUTCOMES:
The rate of organ preservation | 2 years
  Rate of patients who achieve organ preservation
The rate of anus preservation | 2 years
  Rate of patients who achieve anus preservation
pCR rate | 2 years
  Rate of pCR patients after surgery
Disease free survival(DFS) | 2 years
  DFS was defined as the duration from the date of randomization to the date of the first recurrence (local, distant, or mixed) or death.
overall survival(OS) | 2 years
  OS was calculated from the date of randomization.
Quality of life | 2 years
  The QoL was assessed by EORTC QOL Core Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD would be available upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 2 years

REFERENCES:
- [Derived] Zhou L, Yu G, Wen R, Jia H, Zhang T, Peng Z, Fan H, Pan A, Yu Y, Zhu X, Gong H, Gao X, Lou Z, Zhang W. Neoadjuvant chemoradiation therapy combined with immunotherapy for microsatellite stable ultra-low rectal cancer (CHOICE II): study protocol of a multicentre prospective randomised clinical trial. BMJ Open. 2023 Sep 13;13(9):e069793. doi: 10.1136/bmjopen-2022-069793. PMID 37709314